CLINICAL TRIAL: NCT04799496
Title: Regulatory Post-Marketing Surveillance Study (Usage Results Study) of Kynteles Injection (Vedolizumab) for the Approved Indications in South Korea
Brief Title: A Study of Kynteles Injection (Vedolizumab) in Adults With Moderate to Severe Ulcerative Colitis or Crohn's Disease or Chronic Pouchitis
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-4023
Record Dates: First submitted 2021-03-15; First posted 2021-03-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kynteles Injection (Vedolizumab): Participants with moderately to severely active UC and CD, who have had an inadequate response with, lost response to, or were intolerant to either conventional therapy or a tumor necrosis factor-alpha (TNF-α) antagonist or participants with pouchitis, who have undergone proctocolectomy and IPAA for UC, and have had an inadequate response with, or lost response to antibiotic therapy and have initiated Kynteles injection (Vedolizumab) treatment in a routine clinical practical setting in South Korea, will be observed prospectively.

SUMMARY:
In this study, participants with ulcerative colitis or Crohn's disease or pouchitis will be treated with Kynteles injection (Vedolizumab) according to their clinic's standard practice.

The main aim of the study is to check for side effects from treatment with Kynteles injection (Vedolizumab). Another aim is to learn how many participants have improved symptoms after treatment with Kynteles injection (Vedolizumab).

DETAILED DESCRIPTION:
This is a non-interventional, prospective, post-marketing study of participants with inflammatory bowel disease (IBD) (ulcerative colitis (UC) or Crohn's disease (CD)), who have had an inadequate response with, lost response to, or were intolerant to conventional therapy or an TNF-alpha antagonist or participants with pouchitis, who have undergone proctocolectomy and ileal pouch anal anastomosis (IPAA) for UC, and have had an inadequate response with, or lost response to antibiotic therapy. This study will evaluate the safety and effectiveness of Kynteles injection (Vedolizumab) in a routine clinical practice setting under real world conditions.

This study will enroll approximately 600 participants. The data will be prospectively collected, at the centers from routinely scheduled follow-up visits and recorded into electronic case report forms (e-CRFs).

This multi-center trial will be conducted in South Korea. The overall time for data collection in the study will be approximately 6 years.

ELIGIBILITY:
Inclusion Criteria:

1. With moderately to severely active UC and CD, who have had an inadequate response with, lost response to, or were intolerant to either conventional therapy or a TNF-α antagonist
2. With moderately to severely active chronic pouchitis, who have undergone proctocolectomy and IPAA for UC, and have had an inadequate response with, or lost response to antibiotic therapy.

Exclusion Criteria:

1. With hypersensitivity such as dyspnea, bronchospasm, urticaria, flushing and increased heart rate to the Kynteles Injection (Vedolizumab) or to any of its excipients
2. With active severe infections such as tuberculosis, cytomegalovirus, sepsis, listeriosis and opportunistic infections such as progressive multifocal leukoencephalopathy (PML)
3. Treated with Kynteles Injection (Vedolizumab) outside of the locally approved label in South Korea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll moderately to severely active UC and CD, who have had an inadequate response with, lost response to, or were intolerant to either conventional therapy or a TNF-α antagonist or pouchitis, who have undergone proctocolectomy and IPAA for UC, and have had an inadequate response with, or lost response to antibiotic therapy.
Sampling Method: Probability Sample
Enrollment: 688 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Serious Adverse Events (SAEs) | Baseline up to 56 weeks
Percentage of Participants With Adverse Drug Reactions (ADRs) | Baseline up to 56 weeks
Percentage of Participants With Serious Adverse Drug Reactions (SADRs) | Baseline up to 56 weeks
Percentage of Participants With Adverse Events of Special Interest (AESIs) | Baseline up to 56 weeks
Percentage of Participants With Unexpected Adverse Events (AEs) | Baseline up to 56 weeks
Percentage of Participants With Unexpected ADRs | Baseline up to 56 weeks

SECONDARY OUTCOMES:
Percentage of Participants With Clinical Response | Baseline up to 56 weeks
  Clinical response: reduction of Mayo score of >=3 points and >=30 percent (%) from baseline score, with an accompanying decrease in rectal bleeding sub-score >=1 point/an absolute rectal bleeding sub-score of <=1 point in UC participants; and reduction of Crohn's Disease Activity Index (CDAI) score >=70 points from baseline score in CD participants. Mayo score consists of 4 variables: stool frequency, rectal bleeding, physician rating of disease activity, and endoscopic findings. Each graded from 0-3. Total score range of 0-12. Higher scores indicating more severity. CDAI assesses CD based on clinical signs such as number of liquid stools, intensity of abdominal pain, general wellbeing (subjective), and presence of complications, use of antidiarrheal, presence of abdominal mass, physical examination and hematocrit (objective). CDAI score is equal to sum of weighted scores for subjective and objective items. Total score ranged from 0-600 points. Higher score indicating more severity.
Percentage of Participants With Clinical Remission | Baseline up to 56 weeks
  Clinical remission: Mayo score <=2; no individual sub-score greater than (>) 1 point in UC; CDAI score <150 points in CD; and Modified Pouchitis Disease Activity Index (mPDAI) score <5 and reduction in overall score by greater than or equal to (>=) 2 points from baseline score in pouchitis. Mayo score consists of 4 variables: stool frequency, rectal bleeding, physician rating of disease activity, endoscopic findings. Each graded from 0-3. Total score range: 0-12. Higher scores-more severity. CDAI assesses CD based on clinical signs-number of liquid stools, intensity of abdominal pain, general wellbeing (subjective), and presence of complications, use of antidiarrheal, presence of abdominal mass, physical examination, hematocrit (objective). CDAI score: sum of weighted scores for subjective and objective items. Total score:0-600 points. Higher score-more severity. mPDAI score ranges from 0-12 where <5=quiescent; 5-8=moderately active; 9-12=severely active disease.
Percentage of Participants With Mucosal Healing | Baseline up to 56 weeks
  Mucosal healing is defined as: the Mayo endoscopic sub-score of less than or equal to (<=) 1 point in the UC participants; and Crohn's Disease Endoscopic Index of Severity (CDEIS) score less than (<) 3.5 points in the CD participants. Mayo score consists of 4 variables: stool frequency, rectal bleeding, physician rating of disease activity, and endoscopic findings. Each graded from 0-3. Total score range of 0-12. Higher scores indicating more severity. CDEIS is an index of determining the severity of CD. The CDEIS considers rectum, sigmoid and left colon, transverse colon, right colon, ileum in terms of: deep ulcerations, superficial ulcerations, surface involved by disease and ulcerated surface measured. The presence of ulcerate and non-ulcerated stenosis will be recorded in each segment. Scale ranges from 0-44 with a higher score indicating greater severity of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (43):
- South Korea (43):
  - Soon Chunhyang University Hospital Bucheon, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Good Gang-An Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Chungbuk National University Hospital, Cheongju-si
  - Hallym Univ. Medical Center, Chuncheon
  - Kangwon National University Hospital, Chuncheon
  - Daegu Patima Hospital, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Koo Hospital, Daegu
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Chosun University Hospital, Gwangju
  - Inje University Ilsan Paik Hospital, Gyeonggi-do
  - Hanyang University Medical Center, Gyeonggi-do
  - The Catholic University of Korea, Bucheon ST. Marys Hospital, Gyeonggi-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - DongGuk University International Hospital, Ilsan
  - Ilsan Paik Hospital, Ilsan
  - Jeonbuk National University Hospital, Jeonju
  - CHA University Bundang Medical Center, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - Inje University Sanggye Paik Hospital, Seoul
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - KyungHee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Seoul
  - Kyunghee University Hospital at Gangdong, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St.Mary's Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ulsan university Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/605cd562eb9d7e001f5bc69f